CLINICAL TRIAL: NCT05077319
Title: Characteristics and Outcome of Patients With COVID-19 Associated Respiratory Failure Treated in South Tyrol, Italy
Brief Title: Characteristics and Outcome of Patients With COVID-19 in ICUs in South Tyrol
Status: Completed | Type: Observational
Sponsor: Institute of Mountain Emergency Medicine (Other)
Collaborators: Azienda Sanitaria dell'Alto Adige (Other)
Responsible Party: Principal Investigator, Simon Rauch, Senior researcher; MD, PhD, Institute of Mountain Emergency Medicine
Other Study IDs: 1
Record Dates: First submitted 2021-10-04; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; COVID-19 Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators retrospectively investigate the epidemiology, clinical characteristics and therapeutic interventions of patients with COVID-19 associated respiratory failure admitted to the intensive care units in South Tyrol, Italy.

DETAILED DESCRIPTION:
In this observational, retrospective study the epidemiology, characteristics, therapeutic interventions and outcome of patients with COVID-19 associated respiratory failure admitted to the intensive care units in South Tyrol, Italy, are assessed. Data extracted from the medical patients' records include type and duration of respiratory support (high-flow nasal oxygen, non-invasive ventilation, invasive ventilation), need for tracheostomy, vasopressor needs, antibiotic therapy, corticosteroid treatment, laboratory values (interleukin-6, C-reactive protein, procalcitonin, D-dimer, lymphocyte count), lengths of stay in the ICU and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the intensive care units in South Tyrol due to COVID-19 associated respiratory failure

Exclusion Criteria:

* SARS-CoV-2 patients admitted to the intensive care units in South Tyrol for other pathologies (i.e., not respiratory failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care units in South Tyrol due to COVID-19 associated respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Mortality | Through study completion, an average of 1 year
  Mortality (dead/alive) at discharge from the ICU is defined as primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rauch, MD, PhD, Principal Investigator — Institute of Mountain Emergency Medicine
Locations (1):
- Eurac research, Bolzano, Italy